CLINICAL TRIAL: NCT01919918
Title: Muscle Afferent Feedback Effects in Patients With Heart Failure: The Development of Central Fatigue
Brief Title: Muscle Afferent Feedback Effects in Patients With Heart Failure
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Markus Amann, PhD, University of Utah
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 62914
Record Dates: First submitted 2013-07-29; First posted 2013-08-09 (Estimated); Last update posted 2018-01-08 (Actual); Status verified 2018-01

CONDITIONS: Chronic Heart Failure
MeSH Terms: interventions — Muscle Contraction; Adenosine Triphosphate; Lactic Acid; Protons

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Heart Failure Patients (Other): Patients with heart failure will undergo intervention of muscle contraction with metabolite solution administration. Maximal voluntary muscle contraction exercise with varying metabolite solution administration of adenosine triphosphate, lactate, and protons with phosphate buffer.
  Interventions: Drug: Muscle Contraction with Metabolite Solution Administration
- Control Participants (Other): Healthy control participants will undergo intervention of muscle contraction with metabolite solution administration. Maximal voluntary muscle contraction exercise with varying metabolite solution administration of adenosine triphosphate, lactate, and protons with phosphate buffer.
  Interventions: Drug: Muscle Contraction with Metabolite Solution Administration

INTERVENTIONS:
Drug: Muscle Contraction with Metabolite Solution Administration — Participants will perform maximal elbow flexor or knee extensor contractions before and after administration of metabolite solutions of pH 7.2, pH 7.0 and pH 6.6
  Other Names: adenosine triphosphate, lactate, and protons with phosphate buffer

SUMMARY:
The purpose of the study is to find out more about the mechanism by which neural feedback from the working muscle affects the development of central fatigue during exercise. Subjects with chronic heart failure (HF) and healthy subject counterparts will be tested to determine the mechanisms accounting for the premature fatigue characterizing HF patients during physical activity.

DETAILED DESCRIPTION:
A substantial part in limiting exercise and/or physical activity in humans results from the development of peripheral and central fatigue during physical activity. Peripheral fatigue comprises biochemical changes within the metabolic milieu of the working muscle leading to an attenuated response to neural excitation, while central fatigue comprises a failure of the central nervous system to drive motoneurons.

Patients with HF have overactive group III/IV muscle afferents and an exaggerated development of central fatigue during physical activity that is not explained by their reduced physical conditioning or cardiac insufficiency caused by their failing heart. The exact mechanisms accounting for the exaggerated central fatigue in HF remains elusive, however, the development of central fatigue during exercise has recently been linked to signaling by group III/IV muscle afferents. This makes the heightened neural feedback in HF a likely candidate for these patients' increased susceptibility to central fatigue.

Lower pH, increased lactate and increased adenosine triphosphate has been shown to activate group III/IV afferents in a physiological manner and thus induce, in a rested and unfatigued muscle, the intramuscular milieu associated with moderate to heavy exercise. The objective of this study is to quantitate and compare the sensitivity of group III/IV afferents and associated effects on central fatigue in HF patients and healthy controls when skeletal muscle is subject to controlled lower pH, increased lactate and increased adenosine triphosphate.

ELIGIBILITY:
Heart Failure Inclusion Criteria:

* Subjects with a history of stable cardiomyopathy (ischemic and non-ischemic, greater than 1 year duration, ages 20-79 years)
* New York Heart Association class I through IV symptoms
* Left ventricular ejection fraction less than 35 percent (heart failure patients with reduced left ventricular ejection fraction) or greater than 50 percent (heart failure patients with preserved left ventricular ejection fraction)
* Sedentary, no regular physical activity for at least 6 months prior
* Post-menopausal for at least 2 years and follicle stimulating hormone greater than 40

Heart Failure Exclusion Criteria:

* Patients with atrial fibrillation or heart failure believed to be secondary to atrial fibrillation
* Morbidly obese patients with a body mass index greater than 35
* Patients with uncontrolled hypertension, greater than 160/100
* Anemia with a hemoglobin less than 9
* Severe renal insufficiency (creatinine clearance less than 30 by the Cockcroft-Gault formula)
* Patients with significant non-cardiac comorbidities
* Orthopedic limitations that would prohibit them from performing the elbow-flexor exercise
* Current smoker or smoking history of 15 packs or more per year
* Women currently taking hormone replacement therapy

Healthy Control Inclusion Criteria:

* Ages 20-75 years
* Sedentary, no regular physical activity for at least 6 months prior
* Post-menopausal for at least 2 years and follicle stimulating hormone greater than 40

Healthy Control Exclusion Criteria:

* History of cardiovascular related abnormalities or pulmonary abnormalities
* Morbidly obese patients with a body mass index greater than 35
* Patients with uncontrolled hypertension, greater than 160/100
* Anemia with a hemoglobin less than 9
* Orthopedic limitations that would prohibit them from performing the elbow-flexor exercise
* Current smoker or smoking history of 15 packs or more per year
* Women currently taking hormone replacement therapy

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2013-09; Primary Completion 2018-01-03 (Actual); Study Completion 2018-01-03 (Actual)

PRIMARY OUTCOMES:
Elbow Flexor Maximal Voluntary Contraction in newton-meters | 2 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Markus Amann, PhD, Principal Investigator — University of Utah
Locations (2):
- United States (2):
  - George E Wahlen Vetern Affairs Medical Center, Salt Lake City, Utah
  - Veterans Affairs Salt Lake City Heath Care System, Salt Lake City, Utah